CLINICAL TRIAL: NCT05284058
Title: Impact of Preoperative Myocardial Fibrosis Related to Mitral Valve Prolapse on Postoperative Left Ventricular Remodeling
Acronym: IMPARED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_1210; ID-RCB (Other: 2021-A02902-39)
Record Dates: First submitted 2022-02-25; First posted 2022-03-17 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Regurgitation, Mitral
Keywords: Mitral Regurgitation; Myocardial Fibrosis; Surgical Mitral Valve Repair; Cardiac Magnetic Resonance Imaging
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Magnetic Resonance Imaging (Experimental): All patients who are candidates for surgical mitral valve repair through minimally-invasive access according to the standard of care will be considered for inclusion in this clinical study. All patients will undergo cardiac Magnetic Resonance Imaging (MRI) exam before the surgery, as well as at 3 months follow-up.
  Interventions: Other: Cardiac Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Cardiac Magnetic Resonance Imaging (MRI) — Patients will undergo 2 MRI exams: 1 MRI before surgical intervention (maximum 21 days before) and 1 MRI three months after surgery (+/- 14 days), with intravenous administration of gadolinium.

SUMMARY:
Primary mitral regurgitation (MR) is the most common valvular disease in western countries. The MR mechanism is often related to a mitral valve prolapse (MVP) defined as a single or bi-leaflet prolapse of at least 2 mm beyond the long-axis mitral annular plane.

In recent years, several studies have identified a subtype of MVP patients at higher risk of ventricular arrhythmias (VA) and sudden cardiac death (SCD). The presence of regional myocardial replacement fibrosis (RMRF) has been shown as a risk marker of arrhythmic events (VA and SCD) in patients with MVP. RMRF can be identified using cardiac magnetic resonance (CMR) imaging with late gadolinium enhancement (LGE+). In these patients, fibrosis was found in the basal inferolateral myocardium and at the level of papillary muscles (PMs). This fibrosis is developed beyond the volume overload related to the MVP. It is probably linked to the mechanical stretch acting upon the valve and the neighboring left ventricle (LV) myocardium. RMRF is associated with a high degree of MR, with specific features of mitral valve apparatus (bi-leaflet prolapse with marked leaflet redundancy, mitral annulus abnormalities (i.e. Mitral-Annular Disjunction)), and more dilated LV. It is also independently associated with the occurrence of cardiovascular events.

Mitral valve repair (MVr) is the gold standard treatment for primary Mitral Regurgitation. Very little data concerning the impact of preoperative RMRF on mitral valve surgery outcomes is available, and the impact of myocardial fibrosis on the postoperative left ventricle remodeling has not been studied so far.

No previous study compares preoperative and postoperative fibrosis evolution. Thus, no data exists regarding the postoperative evolution of this fibrosis and its relationship with ventricular arrhythmic risk after valve surgery. Small observational studies have suggested that mitral valve surgery did not reduce the risk of ventricular arrhythmias in patients with bileaflet MVP.

Finally, the mechanisms involved in the development of regional myocardial replacement fibrosis within the left ventricle myocardium during the natural history of MVP cannot be understood with current standard medical imaging tools. Numerical simulation technologies provide an innovative and in-vivo approach to assess the physical and pathological mechanisms causing this fibrosis. They can also be used to assess the changes in mitral valve and myocardium dynamics after surgical mitral valve repair procedures.

A large consortium, involving physicians and scientists, has been created to address these questions to fulfil our objectives over a 4 year period (SIMR project).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old)
* Patients candidate for mitral valve repair after validation by the local Heart-Team

  * Severe symptomatic primary Mitral Regurgitation (MR), due to:
  * Posterior or bileaflet prolapse, with
  * Criteria of advance disease (i.e. existence of fibrosis):
* Effective Regurgitant Orifice Area (EROA) > 35 mm2 - Regurgitant volume > 45 mL
* Left ventricular end-diastolic diameter >55 mm
* Left atrium volume index >60 mL/m2
* Pulmonary artery systolic pressure > 30mmHg
* Patients who have provided written informed consent to participate in the study.
* Patients affiliated with a social health insurance.

Exclusion Criteria:

* Patients with contraindication for mitral valve repair, including:

  * Patients with secondary MR; and
  * Calcified leaflets segments.
* Patients with contraindication for a minimally invasive approach including:

  * Previous heart surgery;
  * Previous right lung surgery; or
  * Vascular access contraindications.
* Patients with contraindication for CMR imaging:

  * Patients without sinus rhythm
  * Regular MRI contraindications (e.g. a claustrophobia, a pacemaker, defibrillator or metallic (ferromagnetic) body, a known allergy to gadolinium)
  * Contraindication for Gadolinium infusion: glomerular filtration rate (GFR) <30 ml / min
* Patients unable to understand the purpose of the study
* Patients participating in another trial that would interfere with this study
* Female patients who are pregnant, lactating or women of child-bearing potential without highly effective methods of contraception
* Patients under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Evolution of regional myocardial replacement fibrosis after surgery | at 3 months after surgery
  Evolution of fibrosis mass within the left ventricle myocardium (assessed as Regional late gadolinium enhancement) on cardiac magnetic resonance (CMR) imaging at 3 months after surgery.

SECONDARY OUTCOMES:
Left ventricular volumes | day 0
  Left ventricular volumes assessed by Cardiac Magnetic Resonance Imaging (MRI)
Left ventricular volumes | at 3 months after surgery
  Left ventricular volumes assessed by Cardiac Magnetic Resonance Imaging (MRI)
left ventricular ejection fraction | day 0
  Left ventricular function quantification is assessed by left ventricular ejection fraction in %. by Cardiac Magnetic Resonance Imaging (MRI)
left ventricular ejection fraction | at 3 months after surgery
  Left ventricular function quantification is assessed by left ventricular ejection fraction in %. by Cardiac Magnetic Resonance Imaging (MRI
Extracellular volume | day 0
  Extracellular volume is assessed by Cardiac Magnetic Resonance Imaging (MRI)
Extracellular volume | 3 months after surgery
  Extracellular volume is assessed by Cardiac Magnetic Resonance Imaging (MRI)
Mitral Regurgitation (MR) residual assessment | day 0
  Residual MR is assessed by Cardiac Magnetic Resonance Imaging (MRI)
Mitral Regurgitation (MR) residual assessment | at 3 months after surgery
  Residual MR is assessed by Cardiac Magnetic Resonance Imaging (MRI)
Number of adverse events (AEs) | up to 12 months
  Post-operative safety is assessed by occurrence of adverse events (AEs) and serious adverse events (SAEs) at each of the follow-up times
Number of serious adverse events (SAEs) | up to 12 months
  Post-operative safety is assessed by occurrence of adverse events (AEs) and serious adverse events (SAEs) at each of the follow-up times
New York Heart Association (NYHA) score | at day 0
  Change in functional evaluation is assessed by NYHA functional classification of heart failure. It is based on symptom severity and the amount of exertion needed to provoke symptoms. NYHA heart failure classes are as follows : Class I No limitation of physical activity, Class II Slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest, Class III Marked limitation of physical activity, in which less-than-ordinary activity results in fatigue, palpitation, or dyspnea; the person is comfortable at rest and Class IV Inability to carry on any physical activity without discomfort but also symptoms of heart failure at rest, with increased discomfort if any physical activity is undertaken.
New York Heart Association (NYHA) score | at discharge from hospital (day 15)
  Change in functional evaluation is assessed by NYHA functional classification of heart failure. It is based on symptom severity and the amount of exertion needed to provoke symptoms. NYHA heart failure classes are as follows : Class I No limitation of physical activity, Class II Slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest, Class III Marked limitation of physical activity, in which less-than-ordinary activity results in fatigue, palpitation, or dyspnea; the person is comfortable at rest and Class IV Inability to carry on any physical activity without discomfort but also symptoms of heart failure at rest, with increased discomfort if any physical activity is undertaken.
New York Heart Association (NYHA) score | at 1 month after surgery
  Change in functional evaluation is assessed by NYHA functional classification of heart failure. It is based on symptom severity and the amount of exertion needed to provoke symptoms. NYHA heart failure classes are as follows : Class I No limitation of physical activity, Class II Slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest, Class III Marked limitation of physical activity, in which less-than-ordinary activity results in fatigue, palpitation, or dyspnea; the person is comfortable at rest and Class IV Inability to carry on any physical activity without discomfort but also symptoms of heart failure at rest, with increased discomfort if any physical activity is undertaken.
New York Heart Association (NYHA) score | at 3 months after surgery
  Change in functional evaluation is assessed by NYHA functional classification of heart failure. It is based on symptom severity and the amount of exertion needed to provoke symptoms. NYHA heart failure classes are as follows : Class I No limitation of physical activity, Class II Slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest, Class III Marked limitation of physical activity, in which less-than-ordinary activity results in fatigue, palpitation, or dyspnea; the person is comfortable at rest and Class IV Inability to carry on any physical activity without discomfort but also symptoms of heart failure at rest, with increased discomfort if any physical activity is undertaken.
New York Heart Association (NYHA) score | at 12 months after surgery
  Change in functional evaluation is assessed by NYHA functional classification of heart failure. It is based on symptom severity and the amount of exertion needed to provoke symptoms. NYHA heart failure classes are as follows : Class I No limitation of physical activity, Class II Slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest, Class III Marked limitation of physical activity, in which less-than-ordinary activity results in fatigue, palpitation, or dyspnea; the person is comfortable at rest and Class IV Inability to carry on any physical activity without discomfort but also symptoms of heart failure at rest, with increased discomfort if any physical activity is undertaken.
The 3-level version of EQ-5D (EQ-5D-3L) health status score (quality of life score) | at day 0
  The EQ-5D-3L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
The 3-level version of EQ-5D (EQ-5D-3L) health status score (quality of life score) | at discharge from hospital (day 15)
  The EQ-5D-3L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
The 3-level version of EQ-5D (EQ-5D-3L) health status score (quality of life score) | at 1 month after surgery
  The EQ-5D-3L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
The 3-level version of EQ-5D (EQ-5D-3L) health status score (quality of life score) | at 3 months after surgery
  The EQ-5D-3L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
The 3-level version of EQ-5D (EQ-5D-3L) health status score (quality of life score) | at 12 months after surgery
  The EQ-5D-3L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
end-diastolic diameter in mm | at day 0
  Left ventricular dimension assessed by transthoracic echocardiographic exam
end-systolic diameter in mm | at day 0
  Left ventricular dimension assessed by transthoracic echocardiographic exam
Left ventricular volume | at day 0
  assessed by transthoracic echocardiographic exam
end-diastolic diameter in mm | at discharge from hospital (day 15)
  Left ventricular dimension assessed by transthoracic echocardiographic exam
end-systolic diameter in mm | at discharge from hospital (day 15)
  Left ventricular dimension assessed by transthoracic echocardiographic exam
Left ventricular volume | at discharge from hospital (day 15)
  assessed by transthoracic echocardiographic exam
Left ventricular volume | at 1 month after surgery
  assessed by transthoracic echocardiographic exam
end-diastolic diameter in mm | at 1 month after surgery
  Left ventricular dimension assessed by transthoracic echocardiographic exam
end-systolic diameter in mm | at 1 month after surgery
  Left ventricular dimension assessed by transthoracic echocardiographic exam
Left ventricular volume | at 12 months after surgery
  assessed by transthoracic echocardiographic exam
end-diastolic diameter in mm | at 12 months after surgery
  Left ventricular dimension assessed by transthoracic echocardiographic exam
end-systolic diameter in mm | at 12 months after surgery
  Left ventricular dimension assessed by transthoracic echocardiographic exam
Left atrium volume | at day 0
  Left atrium volume are assessed by transthoracic echocardiographic exam
Left atrium volume | at discharge from hospital (day 15)
  Left atrium volume are assessed by transthoracic echocardiographic exam
Left atrium volume | at 1 month after surgery
  Left atrium volume are assessed by transthoracic echocardiographic exam
Left atrium volume | at 12 months after surgery
  Left atrium volume are assessed by transthoracic echocardiographic exam
area | at day 0
  area assessed by transthoracic echocardiographic exam
area | at discharge from hospital (day 15)
  area assessed by transthoracic echocardiographic exam
area | at 1 month after surgery
  area assessed by transthoracic echocardiographic exam
area | at 12 months after surgery
  area assessed by transthoracic echocardiographic exam
Mitral annulus diameter | at day 0
  Mitral annulus diameter is assessed by transthoracic echocardiographic exam
Mitral annulus diameter | at discharge from hospital (day 15)
  Mitral annulus diameter is assessed by transthoracic echocardiographic exam
Mitral annulus diameter | at 1 month after surgery
  Mitral annulus diameter is assessed by transthoracic echocardiographic exam
Mitral annulus diameter | at 12 months after surgery
  Mitral annulus diameter is assessed by transthoracic echocardiographic exam
Mitral Regurgitation (MR) residual assessment | at day 0
  Residual MR is assessed by transthoracic echocardiographic exam
Mitral Regurgitation (MR) residual assessment | at discharge from hospital (day 15)
  Residual MR is assessed by transthoracic echocardiographic exam
Mitral Regurgitation (MR) residual assessment | at 1 month after surgery
  Residual MR is assessed by transthoracic echocardiographic exam
Mitral Regurgitation (MR) residual assessment | at 12 months after surgery
  Residual MR is assessed by transthoracic echocardiographic exam

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pneumologique et Cardiovasculaire Louis Pradel - Hospices Civils de Lyon - Groupement Hospitalier Est, Bron, France